CLINICAL TRIAL: NCT05329181
Title: Integrated Cognitive Behavioral Treatment for Substance Use and Depressive Symptoms: A Homeless Case Series and Feasibility Study
Brief Title: Integrated Cognitive Behavioral Treatment for Substance Use and Depressive Symptoms: a Homeless Case Series
Acronym: INTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Ersta Diakoni (Other)
Responsible Party: Principal Investigator, Brjann Ljotsson, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTER
Record Dates: First submitted 2022-03-21; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated cognitive behavioral therapy adapted for homeless individuals (Other): Four homeless individuals enrolled in the Treatment First program (a social services program where treatment is offered in conjunction with temporary transitional housing), who had access to stable and sober housing milieus, received the integrated cognitive behavioral treatment.
  Interventions: Behavioral: Integrated cognitive behavioral treatment

INTERVENTIONS:
Behavioral: Integrated cognitive behavioral treatment — Integrated cognitive behavioral treatment adapted specifically for homeless individuals and developed to treat substance use and depressive symptoms simultaneously

SUMMARY:
This case series and feasibility trial evaluated a novel integrated cognitive behavioral treatment, which was adapted specifically for homeless individuals and developed to treat substance use and depressive symptoms simultaneously. The integrated cognitive behavioral treatment was delivered among four homeless individuals enrolled in the Treatment First program (a social services program where treatment is offered in conjunction with temporary transitional housing), who had access to stable and sober housing milieus.

DETAILED DESCRIPTION:
All study participants were clients at the social welfare office for the homeless, a specialized unit within the social services in Stockholm, Sweden. The participants were referred to outpatient treatment at Pelarbacken, a specialized primary care center for homeless patients.

The integrated cognitive behavioral treatment was developed as part of a collaborate treatment program between the social welfare office for the homeless and Pelarbacken. Post treatment interviews and individual behavioral analyses of prior patients showed that the far most common reason for alcohol or drug use, was coping with negative affect (46% reported this reason). The integrated cognitive behavioral treatment was developed emanating from the following analysis (1) being homeless often implicates having lost contact with several important life areas, substance use might be the only reinforcing activity left; (2) common reactions are stress and depressive symptoms, and avoidance based strategies such as passivity, isolation, avoidance of social contact, or substance use; (3) when decreasing substance use, a transient approximate 3 month period of increased "depression-like" symptoms occurs, which might lead to lapses or relapses (this period is also called post-acute abstinence, or protracted abstinence). The ICBT (5-15 sessions) was developed to extend over this time period, with the overall aim of participants to (1) access a stable, sober housing milieu, and decrease substance use; (2) learn strategies to cope with negative affect; and (3) learn strategies to cope with life changes, increase activities such as work, social contact, exercise or leisure activities.

Measures were administered at pre treatment, weekly during treatment, after treatment, and at 3-, 6- and 12-month following treatment cessation.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled the Diagnostic and Statistical Manual of Mental Disorders criteria for Alcohol Use Disorder or Substance Use Disorder
* Fulfilled the Swedish criteria for homelessness and had access to "steady housing" (defined as situation 3 or 4 according to Sun et al. [2012])
* Were between 16-65 years old
* Were able to read and write Swedish and were able to carry out treatment, 5-15 sessions together with homework assignments
* Had regular contact with a social worker at the social welfare office for the homeless.

Exclusion Criteria:

* Another primary psychiatric condition (e.g., bipolar disorder, psychosis, suicidal ideation)
* Failure to attend first two treatment sessions
* Other aggravating circumstances, for example violence in close relationships.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
The TimeLine Follow Back | A retrospective 90-day TimeLine Follow Back interview at baseline, and a retrospective 7 days TimeLine Follow Back self-report measure assessed weekly during treatment sessions (up to 15 sessions/weeks).
  The TimeLine Follow Back, a retrospective calendar instrument to assess days and quantity of alcohol and drug use, was used as primary measure for substance use. The TimeLine Follow Back have been found to have good psychometric properties in a homeless population (Sacks et al., 2003). Number of units (alcohol or drug use) per week were reported as means per week, during baseline and treatment. The TimeLine Follow Back was not administered at follow up.

SECONDARY OUTCOMES:
The Patient Health Questionnaire | 1 week
  The Patient Health Questionnaire is a 9-item self-report measure (score range 0-27) that assesses depression severity with the following cut-off categories: None-minimal (0-4), mild (5-9), moderate (10-14), moderately-severe (15-19), severe (20-27).
The Generalized Anxiety Questionnaire | 2 weeks
  The Generalized Anxiety Questionnaire is a 7 item self- report measure (score range 0-21) to assess anxiety, with the following cut-off categories: Mild (5-9), moderate (10-14), severe (15-21).
The Alcohol Use Disorders Identification Test | 1 year
  The Alcohol Use Disorders Identification Test is a 10 item self-report measure (score range 0-40) that assesses alcohol consumption. A cut-off of 8 and 6, indicates a hazardous and harmful pattern of alcohol consumption for men and women, respectively.
The Drug Use Disorders Identification Test | 1 year
  The Drug Use Disorders Identification Test is a 11 item self-report measure (score range 0-44) to identify and assess non-alcohol drug use patterns. A cut-off score of 6 and 2 indicates problematic drug use for men and women, respectively; and a score of ≥25 indicates heavily dependence on drugs.
Housing status | 1 day
  The degree of homelessness was assessed with the questions "When was the last time that you had a housing of your own?" and "Where did you sleep last night?", with response alternatives based upon the Swedish national definition of homelessness: "Outside"; "At a shelter"; "In a temporary (sober) residential institution", "In a reference-based training or trial apartment", or "In my own apartment (own lease)". In addition, information of the participants' housing status was collected from the registers of the social welfare office for the homeless at baseline and follow up.
The Credibility/Expectancy Questionnaire | 1 day
  Treatment credibility and expectancy was measured with the Credibility/Expectancy Questionnaire (score ranges credibility 1-19, and expectancy 0-100%, respectively). Higher scores indicate higher treatment credibility/expectancy.
The Client Satisfaction Questionnaire | 1 day
  Treatment satisfaction was measured with the Client Satisfaction Questionnaire (score range 8-32). Higher scores indicate higher treatment satisfaction.
Adverse events | Through study completion, 1 year
  The participants reported adverse events using a self-report measure adapted for psychological treatment. The adverse events measure does not include a total score or a score range, instead each adverse event experienced during treatment is reported. For each adverse event reported participant also rated the discomfort caused by the event when it occurred, as well as residual discomfort (level of discomfort at the time of assessment). Each adverse event reported is rated between 0 ("did not affect me at all") and 3 ("affected me very negatively").

IPD SHARING:
Plan to Share IPD: No
Data is not possible to share du to integrity reasons, as the study participants were patients.

REFERENCES:
- [Derived] Molander O, Bjureberg J, Sahlin H, Beijer U, Hellner C, Ljotsson B. Integrated cognitive behavioral treatment for substance use and depressive symptoms: a homeless case series and feasibility study. Pilot Feasibility Stud. 2023 May 5;9(1):76. doi: 10.1186/s40814-023-01305-2. PMID 37147667